CLINICAL TRIAL: NCT01478685
Title: A Phase 1 Study of CC-486 as a Single Agent and in Combination With Carboplatin or ABI-007 in Subjects With Relapsed or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZA-ST-001
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Urinary Bladder Neoplasms; Carcinoma, Transitional Cell; Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Pancreatic Ductal; Tumor Virus Infections
Keywords: Relapsed or Refractory Solid Tumors
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell; Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Pancreatic Ductal; Tumor Virus Infections; Recurrence | interventions — cc-486; Azacitidine; Carboplatin; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A: CC-486 plus Carboplatin (Experimental): CC-486 will be administered orally at doses between 100-300 mg daily for either 14 or 21 days depending on tolerability. Carboplatin will be given by intravenous (IV) infusion once every 21 Days at a dosage of AUC x 4.
  Interventions: Drug: CC-486; Drug: Carboplatin
- Arm B: CC-486 plus ABI-007 (Experimental): CC-486 will be administered orally at doses between 100-300 mg daily for either 14 or 21 days depending on tolerability
  ABI-007 will be administered by intravenous (IV) infusion on two of every three weeks at a dosage of 100 mg/m^2
  Interventions: Drug: CC-486; Drug: ABI-007
- Arm C: CC-486 (Experimental): CC-486 will be administered orally at doses between 100-300 mg daily for either 14 or 21 days depending on tolerability
  Interventions: Drug: CC-486

INTERVENTIONS:
Drug: CC-486 — CC-486 will be administered orally at doses between 100-300 mg daily for either 14 or 21 days depending on tolerability
  Other Names: Oral Azacitidine
Drug: Carboplatin — Carboplatin will be given by intravenous (IV) infusion once every 21 Days at a dosage of AUC x 4.
  Other Names: Paraplatin
  Arms: Arm A: CC-486 plus Carboplatin
Drug: ABI-007 — ABI-007 will be administered by intravenous (IV) infusion on two of every three weeks at a dosage of 100 mg/m^2
  Other Names: nab-paclitaxel; Abraxane
  Arms: Arm B: CC-486 plus ABI-007

SUMMARY:
The purpose of the study is to evaluate the safety and to define the Maximal Tolerated Dose (MTD) or the Maximal Administered Dose (MAD) of oral azacitidine as a single agent and in combination with carboplatin (CBDCA) or paclitaxel protein bound particles (ABI-007,ABX) in subjects with relapsed or refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, 18 years or older at the time of signing the Informed Consent Document (ICD).
2. Understand and voluntarily sign an ICD prior to any study-related assessments or procedures are conducted.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. With histological or cytological confirmation of advanced unresectable solid tumors, including those who have progressed on (or not been able to tolerate) standard anticancer therapy, or for whom no other effective therapy exists, or for who declines standard therapy.
5. Consent to screening tumor biopsy (for accessible tumors when appropriate [optional in Part 1, mandatory in Part 2]).
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2.
7. The following laboratory values:

   * Absolute neutrophil count (ANC) ≥ 1.5 X 10^9/L
   * Hemoglobin (Hgb) ≥90 g/L
   * Platelets (plt) ≥ 100 x 10^9/L
   * Potassium within normal range, or correctable with supplements;
   * AST and ALT ≤2.5 x Upper Limit Normal (ULN) or ≤5.0 x ULN if liver tumor is present;
   * Serum total bilirubin ≤ 1.5 x ULN
   * Serum creatinine ≤ 1.5 x ULN, or 24-hr clearance ≥ 60ml/min; and
   * Negative serum pregnancy test within 7 days before starting study treatment in females of childbearing potential (FCBP)
8. Females of child-bearing potential {defined as a sexually mature women who

   * has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or,
   * has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time during the preceding 24 consecutive months} must

     * agree to the use of a physician- approved contraceptive method (oral, injectable, or implantable hormonal contraceptive ; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) while on oral azacitidine and for 3 months following the last dose of study medication; and
     * have a negative serum pregnancy test during screening
9. Male subjects with female partner of childbearing potential must agree to the use of a physician-approved contraceptive method throughout the course of the study to avoid fathering a child during the course of the study and for 6 months following the last dose of oral azacitidine.

The criteria below are in addition to or supersede the Part 1 inclusion criteria above:

1. With histological or cytological confirmation of relapsed or refractory advanced unresectable solid tumors as listed below for each Arm, including those who have progressed on or were unable to tolerate standard anti-cancer therapy.

   * Arm A: CC-486 plus CBDCA:
   * Relapsed or refractory urothelial carcinoma of the bladder, renal pelvis, ureter, or urethra (mixed histologies are permitted provided a component of urothelial carcinoma is present)
   * Epithelial ovarian, fallopian tube, or primary peritoneal carcinoma
   * Arm B: CC-486 plus ABI-007:
   * NSCLC
   * Pancreatic carcinoma
   * Arm C: CC-486 single agent:
   * Virally-associated tumors - tumor types known to be driven by Epstein-Barr Virus (EBV), Human Papilloma Virus (HPV), and Merkel cell carcinoma of the skin (MC Polomavirus)
   * Nasopharyngeal carcinoma (a minimum of 5 subjects)
   * Cervical carcinoma
   * Anal carcinoma
   * Merkel cell carcinoma (MCC)
   * Note: Hepatitis B virus (HBV) and Hepatitis C virus (HCV)-associated tumors (hepatocellular cancers) are not eligible.
   * Note: Head and neck squamous cell cancers (HNSCC) must have HPV-positive status documented to be eligible
2. Subjects with documented liver metastases must have serum albumin ≥ 3 g/dL;
3. Sites of disease (primary or metastatic) that are, in the opinion of the investigator, accessible for biopsy without undue risk to the subject
4. Consent to tumor biopsy at screening (prior to the first dose of CC-486) and at Cycle 1 Day 15.
5. Measurable disease according to RECIST v1.1.

Exclusion Criteria:

1. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Any condition that confounds the ability to interpret data from the study.
4. Symptomatic central nervous system metastases. Subjects with brain metastases that have been previously treated and are stable for 6 weeks are allowed.
5. Known acute or chronic pancreatitis.
6. Any peripheral neuropathy ≥ NCI CTCAE grade 2.
7. Persistent diarrhea or malabsorption ≥ NCI CTCAE grade 2, despite medical management.
8. Impaired ability to swallow oral medication.
9. Unstable angina, significant cardiac arrythmia, or New York Heart Association (NYHA) class 3 or 4 congestive heart failure.
10. Prior systemic cancer-directed treatments or investigational modalities ≤ 5 half lives or 4 weeks, whichever is shorter, prior to starting study drug or who have not recovered from side effects of such therapy. (except alopecia).
11. Major surgery ≤ 2 weeks prior to starting a study drug or who have not recovered from side effects of such therapy.
12. Pregnant or breast feeding.
13. Known Human Immunodeficiency Virus (HIV) infection.
14. Known chronic hepatitis B or C virus (HBV/HCV) infection, unless this is a comorbidity in subjects with HCV.
15. Liver metastases with serum albumin < 3 g/dL.
16. Other prior cancers within previous 5 years except adequately treated in situ carcinoma cervix, or basal, or squamous carcinoma of the skin.
17. Subjects with > 4 prior systemic chemotherapy regimens will require approval by the Celgene Medical Monitor prior to enrollment. A regimen is defined as >/= 2 cycles of systemic anti-cancer therapy containing 1 or more agents in the following classes: topoisomerase 1 or 2 inhibitors, platinum salts, alkylating agents, tubulin inhibitors, anti-metabolites or vinca alkaloids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2011-11-29 (Actual); Primary Completion 2015-11-17 (Actual); Study Completion 2015-11-17 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 3 years
  An adverse event (AE) is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. Any worsening (i.e., any clinically significant adverse change in the frequency or intensity.

SECONDARY OUTCOMES:
Cmax | Up to 30 days
  Maximum observed concentration in plasma (Cmax)
AUC | Up to 30 days
  Area under the concentration-time curve (AUC)
Tmax | Up to 30 days
  Time to maximum concentration (tmax);
T1/2 | Up to 30 days
  Terminal half-life (t1/2)
CL/F | Up to 30 days
  Apparent total body clearance (CL/F)
Vz/F | Up to 30 days
  Apparent volume of distribution (Vz/F).
DNA Methylation | Up to 30 days
  Change from baseline (Cycle 1 Day 1 pre-dose) in DNA methylation (global and gene-specific assays) in whole blood and tumor tissue (as available in Part 1)
DNMT1 protein levels | Up to 30 days
  Reduction from baseline (Cycle 1 Day 1 predose) in DNMT1 protein levels in tumor tissue (as available in Part 1)
Tumor Response Rate | Up to 3 years
  Response and progression were evaluated using the RECIST 1.1 criteria. Treatment response includes both complete response and partial response.
  * Complete response-disappearance of all lesions
  * Partial response-30% decrease in the sum of diameters of target lesions from baseline
Progression Free Survival | Up to 3 years
  Progression-free survival is defined as the time from first dose of study drug to the start of disease progression or patient death, whichever occurs first.
Duration of Response | Up to 3 years
  Duration of response is defined as progression-free survival in responders, i.e. as the time between the start of a complete response (CR) or partial response (PR) and the start of progressive disease (PD) or patient death from any cause, whichever occurred first

CONTACTS AND LOCATIONS:
Overall Officials: Gordan Bray, M.D., Ph.D, Study Director — Celgene
Locations (13):
- United States (7):
  - Scottsdale Healthcare Research Institute, Scottsdale, Arizona
  - University of California, San Francisco, San Francisco, California
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Karmanos Cancer Institute, Detroit, Michigan
  - Greenville Hospital, Greenville, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
- France (2):
  - Centre Georges Francois Leclerc, Dijon
  - Institut Curie, Paris
- Netherlands (2):
  - The Netherlands Cancer Instiute Antoni Van Leeuwenhoekziekenhuis, Amsterdam
  - Erasmus Medical Center, Rotterdam
- Spain (2):
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

REFERENCES:
- [Background] LoRusso P, et al. A Phase Ib study of CC-486 (Oral Azacitidine) as a priming agent for carboplatin or NAB-paclitaxel in subjects with relapsed and refractory solid tumors . Presented at 25th AACR-NCI-EORTC Symposium on Molecular Targets and Cancer Therapeutics, October 19-23, 2013, Boston, MA. Abstract No. A120.